CLINICAL TRIAL: NCT03294993
Title: Doppler Ultrasonography Assessed Vascular Changes Before and After Radial Artery Puncture
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Associate proffesor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20170711
Record Dates: First submitted 2017-09-20; First posted 2017-09-27 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Blood Flow Indexes

STUDY DESIGN:
Intervention Model Description: Doppler Ultrasonography Assessed Vascular Changes Before and After Radial Artery Puncture
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound assess group (Experimental): The investigators designed a study to assess whether there were any blood flow indexes change before and after radial artery puncture with doppler ultrasonography
  Interventions: Device: Ultrasound assess

INTERVENTIONS:
Device: Ultrasound assess — The investigators designed a study to assess whether there were any blood flow indexes change before and after radial artery puncture with doppler ultrasonography

SUMMARY:
The investigators designed a study to assess whether there were any blood flow indexes change before and after radial artery puncture with doppler ultrasonography

DETAILED DESCRIPTION:
The investigators designed a study to assess whether there were any blood flow indexes change before and after radial artery puncture with doppler ultrasonography.The indexes include Arterial Diameter,Peak Systolic Velocity,End Diastolic Velocity,Resistive Index,Pulsatility Index,Systolic/End Diastolic Ratio,Time AverageMean Velocity and Blood Flow.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the study if they were ethnic Chinese, between 18 and 65 years old, American Society of Anesthesiologists (ASA) physical status I or II,candidates for general anesthesia undergoing thoracic surgery

Exclusion Criteria:

* Patients were excluded if they do not want to cooperate with the test, had a history of upper extremity arteriosclerosis obliterans or thromboangitis obliterans,had a history of radial artery puncture or coronary artery bypass grafting,had acute vessel trauma,or had been diagnosed with Raynaud' disease,had suffered from mental or neurological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The Change of Peak Systolic Velocity | baseline and 30 minutes after surgery
  The Change of Peak Systolic Velocity before and after surgery

SECONDARY OUTCOMES:
the change of modified Allen test | baseline and 30 minutes after surgery
  the change of modified Allen test before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ma, MD,PhD, Study Chair — Department of Anesthesiology
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided